CLINICAL TRIAL: NCT03060109
Title: Fresh Intravenous Blood Samples for TBI Diagnostic Assay Development With Philips Point of Care System (FIRST DOWN)
Brief Title: Fresh Intravenous Blood Samples for TBI Diagnostic Assay Development With Philips Point of Care System
Acronym: FIRST DOWN
Status: Terminated | Type: Observational
Why Stopped: Diagnostic platform no longer under development; study termination not related to any safety issues
Sponsor: Banyan Biomarkers, Inc (Industry)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: ATO-13
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic brain injury; Head injury
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected traumatic brain injury
  Interventions: Other: Blood draw within 12 hours of injury

INTERVENTIONS:
Other: Blood draw within 12 hours of injury

SUMMARY:
The purpose of this study is to collect fresh whole blood within 12 hours from suspected mild head injury (Glasgow Coma Scale score 13-15) from subjects over the age of 18, to help verify that both UCH-L1 and GFAP can be detected with the Philips Minicare POC diagnostic test platform.

ELIGIBILITY:
Inclusion Criteria:

* The Subject is at least 18 years of age at screening.
* The Subject has presented to a Health Care Facility or Emergency Department with a suspected traumatically induced head injury, as a result of insult to the head from an external force.
* The Subject has a Glasgow Coma Scale score of 13-15 at the time of Informed Consent.
* The venous blood sample is collected no later than 12 hours from the time of head injury.
* The Subject is competent and willing to undergo the Informed Consent process

Exclusion Criteria:

* Participating in any other interventional, therapeutic clinical study (an observational study would be acceptable).
* Time of suspected head injury cannot be determined.
* Venipuncture not feasible (i.e., skin integrity compromised at the venipuncture sites, blood vessel calcification (i.e., IV drug users, advanced atherosclerosis) both upper limbs missing (congenital or amputee)).
* Blood transfusion after head injury, and prior to study blood draw
* Blood donation within 1 week of study enrollment.
* The subject is a female who is pregnant or lactating.
* The Subject is otherwise determined by the Principal Investigator to be an unsuitable candidate for participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Suspected head injury subjects over the age of 18 who present to the HCF or ED within 12 hours from the time of head injury. Subjects who will be permitted into the study include those who will meet all the inclusion criteria and will have none of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2017-09-10 (Actual); Study Completion 2017-09-10 (Actual)

PRIMARY OUTCOMES:
Measurement of biomarkers | 12 hours
  Measurement of UCH-L1 and GFAP using Philips Minicare

CONTACTS AND LOCATIONS:
Locations (4):
- Netherlands (4):
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Haaglanden MC Westeinde, The Hague